CLINICAL TRIAL: NCT03939715
Title: Anterior And Multi-Compartment Vaginal Prolapse Repair Augmented With Decellularized Human Dermal Allograft: A Prospactive, Randomized Controlled, Post Market Study
Brief Title: Surgical Intervention With DermaPure vs Native Tissue in Pelvic Organ Prolapse
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Colorado Pelvic Floor Consultants (Industry)
Collaborators: Tissue Regenix Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1385925-1
Record Dates: First submitted 2019-04-30; First posted 2019-05-07 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- DermaPure (Active Comparator)
  Interventions: Biological: DermaPure®
- Native Tissue (Active Comparator)
  Interventions: Procedure: native tissue

INTERVENTIONS:
Biological: DermaPure® — Surgical intervention using DermaPure®
  Arms: DermaPure
Procedure: native tissue — Surgical intervention using native tissue
  Arms: Native Tissue

SUMMARY:
Comparing FDA-approved DermaPure with patient's own native tissue surgically for diagnosis of pelvic organ prolapse.

DETAILED DESCRIPTION:
The investigator is comparing FDA-approved DermaPure with patient's own native tissue for the repair of pelvic organ prolapse. Please see below for detailed objectives and endpoints for our measuring parameters:

Objectives

Specific Aim #1:

To determine the relative safety and efficacy of anterior and multi-compartment vaginal wall prolapse repair augmented with decellularized human dermal allograft (DermaPure®) versus anterior and multi-compartment repair employing native tissue.

Specific Aim #2:

To evaluate bulge symptoms, quality of life, sexual function, and patient satisfaction

Our hypothesis is that pelvic organ prolapse repair augmented with DermaPure® will provide superior anatomic outcomes as compared to native tissue controls with a non-inferior safety profile.

Endpoints

Safety Endpoint #1:

The relative proportion of allograft, native tissue, and procedure-related SAE's at 12 months.

Safety Endpoint #2:

The relative proportion of allograft, native tissue, and procedure-related AE's of interest at 12 months, which include:

* Vaginal shortening
* Vaginal scarring or banding
* De novo vaginal bleeding
* Atypical vaginal discharge
* Fistula formation
* De novo dyspareunia
* Pelvic pain
* Peri-operative infection
* Vaginal infection
* UTI
* Neuromuscular disorder
* SUI (worsening or de novo)
* UUI (worsening or de novo)
* Difficulty emptying bladder (worsening or de novo)
* Graft exposure (into vagina)
* Graft erosion (into viscus)

Efficacy Endpoint #1:

The proportion of patients in each group at 36 months with prolapse of the target compartment beyond the hymen.

Efficacy Endpoint #2:

The proportion of patients in each group at 36 months with bulge symptoms attributable to the target compartment as determined by PFDI-20 question number 3 ("Does the participant usually have a bulge or something falling out that the participant can see or feel in the vaginal area") answering "yes" and >= 2 (responses of "somewhat", "moderately", or "quite a bit"). (Barber)

Efficacy Endpoint #3:

The proportion of patients in each group at 36 months requiring re-treatment for recurrent prolapse of the target compartment (to include surgery, physical therapy or pessary insertion).

Efficacy Endpoint #4:

Change in quality of life in each group from baseline to 36 months as measured by the PFDI-20 and the PFIQ-7. (Barber)

Efficacy Endpoint #5:

Change in sexual function in each group from baseline to 36 months as measured by the PISQ-IR. (Rogers)

Efficacy Endpoint #6:

Patient satisfaction in each group at 36 months as measured by the SSQ-8. (Haff)

Efficacy Endpoint #7:

Patient impression in each group at 36 months of postoperative improvement by the PGI-I (Srikrishna)

ELIGIBILITY:
Inclusion criteria:

* Subject is female
* Subject is at least 18 years of age
* Subject has prolapse of the anterior compartment beyond the hymen
* Subject reports bulge symptoms as defined in question 3 of the PFDI-20 with a response of 2 or higher ("somewhat", "moderately" or "quite a bit")
* Subject is willing and able to provide informed consent
* Subject is willing and able to comply with the follow-up protocol through 36 months

Exclusion criteria:

* Subject is pregnant or intends to become pregnant during the study
* Subject has untreated severe urogenital atrophy
* Subject has an active or chronic systemic infection including any gynecologic infection, untreated urinary tract infection (UTI), or tissue necrosis
* Subject has a history of pelvic organ cancer (e.g. uterine, ovarian, bladder, or cervical)
* Subject has had prior pelvic radiation therapy
* Subject has taken systemic steroids within the last month, or immunosuppressive or immunomodulatory treatment within the last 3 months (list attached)
* Subject has a history of poor wound healing with or without a diagnosis of connective tissue disease
* Subject has chronic systemic pain that includes the pelvic area or chronic focal pain that involves the pelvis
* Subject has uncontrolled diabetes mellitus (DM) as defined by a hemoglobin A1C < or = to 8% (Underwood, Ata)
* Subject has a known neurologic or medical condition that may effect of currently affects bladder function
* Subject is seeking obliterative vaginal surgery as treatment for pelvic organ prolapse (colpocleisis)
* Subject is not able to conform to the modified dorsal lithotomy position
* Subject is currently participating in or plans to participate in another pelvic organ prolapse related study during this study
* Subject has had previous prolapse repair with synthetic mesh in the anterior compartment
* Subject is planning to undergo a concomitant prolapse repair in a non-target compartment with anything other than native tissue or DermaPure®
* Subject is unable to be treated in the anterior compartment with DermaPure®
* Subject is desirous of a concomitant hysteropexy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-05 (Estimated); Primary Completion 2022-05-05 (Estimated); Study Completion 2022-05-05 (Estimated)

PRIMARY OUTCOMES:
Safety through AE and SAE assessments and percentage of incidences | 3 years
  The relative proportion of allograft, native tissue, and procedure-related SAE's is assessed at 12 months, 24 months, and 36 months.
  The relative proportion of allograft, native tissue, and procedure-related AE's of interest is assessed at 12 months, 24 months, and 36 months which include:
  * Vaginal shortening
  * Vaginal scarring or banding
  * De novo vaginal bleeding
  * Atypical vaginal discharge
  * Fistula formation
  * De novo dyspareunia
  * Pelvic pain
  * Peri-operative infection
  * Vaginal infection
  * UTI
  * Neuromuscular disorder
  * SUI (worsening or de novo)
  * UUI (worsening or de novo)
  * Difficulty emptying bladder (worsening or de novo)
  * Graft exposure (into vagina)
  * Graft erosion (into viscus)
Quality of Life through the administration of questionnaires, analyzed at the end of the study as % of patients that are satisfied or above satisfied | 3 years
  The proportion of patients in each group at 36 months with bulge symptoms attributable to the target compartment as determined by PFDI-20 question number 3 ("Do you usually have a bulge or something falling out that you can see or feel in the vaginal area") answering "yes" and >= 2 (responses of "somewhat", "moderately", or "quite a bit"). (Barber) Change in quality of life in each group from baseline to 36 months as measured by the PFDI-20 and the PFIQ-7. (Barber)

CONTACTS AND LOCATIONS:
Overall Officials: James Lukban, DO, Principal Investigator — Colorado Pelvic Floor Consultants
Locations (1):
- Colorado Pelvic Floor Consultants, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF